CLINICAL TRIAL: NCT05436327
Title: Improving Communication for Cancer Treatment: Addressing Concerns of Older Cancer Patients and Caregivers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-0881; NCI-2022-05359 (Other: NCI-CTRP Clinical Trials Processing Registry)
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Aging; Communication
MeSH Terms: conditions — Neoplasms; Communication | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Geriatric Assessment (GA) (Other): Clinical staff undergo training in GA and are provided with facilitation and support for one year as they implement GA among older adult patients (65+) considering chemotherapy and their care partners/caregivers.
  Interventions: Behavioral: Geriatric Assessment

INTERVENTIONS:
Behavioral: Geriatric Assessment — Clinical staff receive (a) training in GA and workflow management strategies (<60 minutes) at baseline, (b) monthly facilitation and technical support calls (15-30 minutes) for 12 months, and (c) a group-based quarterly call for 12 months. For 12 months, clinical staff implement GA strategies during visits with older adult (65+) patients planning to receive new chemotherapy regimen and their care partners/caregivers.

SUMMARY:
To improve patient-centered outcomes for older patients with cancer considering or receiving chemotherapy and their caregivers. To do this, the project team will (a) establish the effectiveness of GA on communication about age-related concerns, patient and caregiver satisfaction with communication about age-related concerns, quality of life, and patient-reported side effects of chemotherapy; (b) evaluate the success of the implementation strategies on the adoption, reach, and fidelity of implementing the GA in community oncology practices; and (c) identify the resources needed to implement GA and the GA-guided recommendations in community oncology practices for older patients considering or receiving chemotherapy.

DETAILED DESCRIPTION:
Objectives:

* Establish the effectiveness of GA on patient and caregiver satisfaction and communication about age-related concerns for older patients receiving chemotherapy in community oncology practices.
* Evaluate the success of our implementation strategies on the reach, adoption, and fidelity of implementing the GA in community oncology practices.
* Identify the resources needed to implement GA and the GA-guided recommendations in community oncology practices for older patients receiving chemotherapy.

ELIGIBILITY:
Practice Staff Participants

Inclusion Criteria:

* Aged 18 years or older
* A practicing clinician (e.g., oncologist, nurse practitioners, physician assistant, advanced practice nurse, registered nurse, medical assistant) or other practice staff (e.g., administrators and IT)
* Fluent in English (reading and speaking)
* Have access to computer, laptop, tablet, or smart phone

Exclusion Criteria:

* Have plans to leave the practice in six months (e.g., retiring or changing organizations)
* Unable to provide consent

Patient Participants

Inclusion Criteria:

* Aged 65 and older
* Considering a new chemotherapy plan

Exclusion Criteria:

• Have been diagnosed with a health condition that precludes their ability to participate in informed consent or in the intervention (e.g., dementia which limits decision-making capacity).

Care Partner/Caregiver Participants (Care partners can be any partner, spouse, family member, and/or friend that has been identified by the patient and/or clinical team that supports the patient through treatment.)

Inclusion Criteria:

* Aged 18 years and older
* Fluent in English (reading and speaking)
* Have access to computer, laptop, tablet, or smart phone

Exclusion Criteria:

• Unable to provide consent

Inclusion of Special Populations:

Employees. The rationale for including employees is to gain a better understanding of how we can improve cancer care for older patients with cancer receiving chemotherapy. It is possible that some employees may be pregnant women or military personnel. We intend to include these individuals as long as they meet the inclusion and exclusion criteria because this is a clinical improvement project to promote the implementation of the GA in routine clinical practice and should have external validity. These individuals would not be excluded in other clinical improvement projects outside of a research study.

Other special populations. This study will not include other special subject populations (students, Non-English-Speaking Populations, Minors, Human Fetuses; Neonates (infants under 30 days old), prisoners/detainees (wards)) because the purpose of the study is to understand the implementation of the GA in clinical oncology practices and its impact on patients 65+ with cancer and their care partners satisfaction with care, communication about their care, quality of life, and patient (65+) reported toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Reach of Geriatric Assessment (GA) implementation in routine medical practice | monthly over 12 months of implementation, and 6 months after implementation
Reach of Geriatric Assessment (GA) implementation in routine medical practice as measured by applying the reach formula (# people served divided by potential # of people) to the following four metrics: | monthly over 12 months of implementation, and 6 months after implementation
  a) patients per month who received the Geriatric Assessment (GA), b) patients per month who received Geriatric Assessment (GA)-guided recommendations, c) total patients per month age 65+, d) total patients per month who were age 65+ and receiving new chemotherapy or deciding to start chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Marie Lowenstein, PhD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org